CLINICAL TRIAL: NCT00135642
Title: Randomized Double Blind Placebo Controlled Trial of Grass Pollen Immunotherapy Using a Cluster Regime
Brief Title: Grass Pollen Immunotherapy Using a Cluster Regime for Seasonal Rhinitis and Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: ALK-Abelló A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DHRG-CLUSTER
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Hayfever; Subcutaneous Immunotherapy; Grass pollen immunotherapy; Seasonal Allergic Rhinoconjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Blood Specimen Collection

INTERVENTIONS:
Biological: Subcutaneous Alutard SQ grass pollen (Phleum pratense)
Procedure: Venepuncture: 20 ml blood sample taken on 2 separate visits

SUMMARY:
The purpose of this study was to assess the effects of grass pollen immunotherapy on symptoms, bronchial hyperresponsiveness and quality of life in seasonal rhinitis and asthma. Hay fever symptoms and medication use, health-related quality of life, and measurements of non-specific bronchial responsiveness were recorded during the study period.

DETAILED DESCRIPTION:
This was a single centre, randomized, double-blind, placebo-controlled, parallel group study. The main aim of this study was to assess the effects of grass pollen immunotherapy on symptoms, bronchial hyperresponsiveness, and quality of life in seasonal rhinitis and asthma. Forty-four patients with severe summer hay fever (of whom 36 reported seasonal chest symptoms and 28 had seasonal bronchial hyperresponsiveness) participated in a randomised double-blind, placebo-controlled, parallel group study. After symptom monitoring for one summer, participants matched placebo injections (n=22) in a rapid up-dosing cluster regimen for 4 weeks, followed by monthly injections for 2 years. Outcome measures included hay fever symptoms and medication use, health-related quality of life, and measurements of non-specific bronchial responsiveness.

Results: Significant reductions were observed in immunotherapy group compared with the placebo group in hay fever symptoms (49%, 15%: P = 0.1), medication scores (80%, 18%; P=.007), and seasonal chest symptoms (90%, 11%; P < .05). Impairment of overall quality of life (mean score of 7 domains) during the pollen season was less in the immunotherapy group than in the placebo group (median difference [95% CI], 0.8 [0.18-1.5]; P=.05=2]. During the pollen season, there was no change in airway methacholine PC20 (provocation concentration producing a 20% fall in FEV1) in the immunotherapy-treated group (P=5), compared with an almost 3 doubling-dose decrease in the placebo-treated group (P=.5), compared with an almost 3 doubling dose decrease in the placebo-treated group (P=.01, between-group difference). There were no significant local or systemic side effects during the study.

Conclusion: Grass pollen immunotherapy improves quality of life in seasonal allergic rhinitis and reduces seasonal asthma symptoms and bronchial hyperresponsiveness.

Note: Ongoing mechanistic studies and nasal biopsies studies until 2008

ELIGIBILITY:
Inclusion Criteria:

* Male and female 18-60 years of age
* Written informed consent obtained before entering the trial
* A clinical history of grass pollen induced allergic rhinoconjunctivitis of two years or more requiring treatment during the grass pollen season
* A clinical history of severe rhinoconjunctivitis symptoms (interfering with usual daily activities or sleep), which remain troublesome despite treatment with anti-allergic drugs during the grass pollen season
* Positive Skin Prick Test (SPT) response (wheal diameter ≥ 5 mm) to Phleum pratense
* Positive specific IgE against Phleum pratense (≥ IgE Class 2)
* Physical examination with no clinically relevant findings
* If pre-menopausal female of childbearing potential, the subject must test negative on standard urine pregnancy test and must be willing to practice appropriate contraceptive methods for the duration of the trial
* Patients with seasonal asthma only if their baseline methacholine PC20 was greater than 2 mg/mL (normal range > 16 mg/ mL)
* Willingness to comply with this protocol

Exclusion Criteria:

* FEV1 < 70% of predicted value
* A clinical history of symptomatic seasonal allergic rhinitis and/or asthma due to tree pollen or weed pollen adjacent to the start of - and potentially overlapping - the grass pollen season
* A clinical history of significant symptomatic perennial allergic rhinitis and/or asthma caused by an allergen to which the subject is regularly exposed
* A clinical history of significant recurrent acute sinusitis (defined as 2 episodes per year for the last two years all of which required antibiotic treatment) or chronic sinusitis
* At randomisation, current symptoms of, or treatment for, upper respiratory tract infection, acute sinusitis, acute otitis media or other relevant infectious process (serous otitis media is not an exclusion criterion)
* History of emergency visit or admission for asthma in the previous 12 months
* Use of an investigational drug within 30 days prior to screening
* Previous treatment by immunotherapy with grass pollen allergen or any other allergen within the previous 5 years
* History of anaphylaxis, including anaphylactic food allergy, bee venom anaphylaxis, exercise anaphylaxis or drug induced anaphylaxis
* History of angioedema
* Any of the following underlying conditions known or suspected to be present:

  * Cystic fibrosis
  * Malignancy
  * Insulin-dependent diabetes
  * Malabsorption or malnutrition
  * Renal or hepatic insufficiency
  * Chronic infection
  * Drug dependency or alcoholism
  * Ischemic heart disease or angina requiring current daily medication or with any evidence of disease making implementation of the protocol or interpretation of the protocol results difficult or jeopardising the safety of the subject (e.g. clinically significant cardiovascular, serious immunopathologic, immunodeficiency whether acquired or not, hepatic, neurologic, psychiatric, endocrine, or other major systemic disease)
* Immunosuppressive treatment
* History of hypersensitivity to the excipients of the trial medications
* History of allergy, hypersensitivity or intolerance to trial medications or rescue medications
* A mental condition rendering the subject unable to understand the nature, scope and possible consequences of the trial, and/or evidence of an uncooperative attitude
* Unlikely to be able to complete the trial, for any reason, or likely to travel for extended periods of time during the grass pollen season

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44
Dates: Start 1996-02; Study Completion 1998-10

PRIMARY OUTCOMES:
Symptom and medication score recorded by subjects
Adverse events

SECONDARY OUTCOMES:
Rhinoconjunctivitis Quality of Life Questionnaire
Seasonal bronchial hyperresponsiveness
Intradermal allergen challenge

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Durham, Professor, Principal Investigator — Royal Brompton Hospital, NHLI Imperial College London United Kingdom
Locations (1):
- Royal Brompton Hospital, NHLI Imperial College, London, United Kingdom